CLINICAL TRIAL: NCT02014181
Title: Flaxseed Modulates Oxidative Stress and Inflammatory Biomarkers in Stable Patients With Cystic Fibrosis and Healthy Controls
Brief Title: Flaxseed Modulates Inflammation and Oxidative Stress in CF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 815533
Record Dates: First submitted 2013-11-27; First posted 2013-12-18 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2012-04

CONDITIONS: Cystic Fibrosis; Oxidative Stress; Inflammation
Keywords: cystic fibrosis; isoprostanes; 8-oxo-dGuo; oxidative stress; inflammation; flaxseed; enterodiol; enterolactone
MeSH Terms: conditions — Cystic Fibrosis; Inflammation | interventions — Linseed Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Flaxseed (Experimental): 40 grams finely ground flaxseed powder daily for one month in patient with cystic fibrosis
  Interventions: Dietary Supplement: finely ground flaxseed powder

INTERVENTIONS:
Dietary Supplement: finely ground flaxseed powder — 40 grams finely ground flaxseed powder daily for one month to patients with cystic fibrosis
  Other Names: flaxseed; Flax; Linseed oil; SDG; Bene-flax

SUMMARY:
Flaxseed (FS) is a safe and well tolerated supplement with an ability to fight inflammation and oxidative stress - a byproduct of daily stress the human body faces everyday and especially with chronic diseases. Cystic fibrosis (CF) is a genetic disease resulting from a mutation in sodium and chloride transport channels that results in pancreatic insufficiency, chronic sinusitis and chronic lung infections. The investigators hypothesize that chronic inflammation and oxidative stress are a part of the chronic exacerbations that are a part of cystic fibrosis. The investigators believe that flaxseed with its anti-inflammatory and antioxidative properties can help dampen these stressors on the CF lung and potentially result in fewer exacerbations of CF, fewer antibiotics, fewer hospitalizations, and improved well-being.

DETAILED DESCRIPTION:
Ten patients with steady-state cystic fibrosis (CF) - not hospitalized, not on intravenous antibiotics, with stable FEV1 40-100% predicted were enrolled in a four week long pilot study where-in each patient consumed 40 grams of flaxseed each day, in the form of finely ground flaxseed, however they wished. Prior to starting flaxseed, each week, and then four weeks after each patient had finished taking flaxseed, markers of inflammation and oxidative stress, as well as measurements of flaxseed metabolism were collected. F2-isoprostanes, 8-oxo-dGuo, as well as cytokines including IL-6, TNF-a, IFN-g among others were measured to trend flaxseed effects. Enterolignans - enterodiol and enterolactone (products of flaxseed metabolism) were measured each week as well.

ELIGIBILITY:
Inclusion Criteria:

1. Genetic and clinical diagnosis of cystic fibrosis (CF)
2. FEV1 predicted between 40-100%
3. Age 18-64
4. Pancreatic enzyme adherence (or pancreatic sufficiency)
5. Demonstration of continued long-term dedication and follow-up with CF primary care provider

Exclusion Criteria:

1. Prior or planned hospitalization or surgical procedure within one month of enrollment (other than simple dental procedure)
2. An acute pulmonary exacerbation
3. History of bowel resection, inflammatory bowel disease or distal intestinal obstruction syndrome
4. Receiving broad spectrum intravenous antibiotics (other than maintenance azithromycin, inhaled tobramycin, or inhaled aztreonam within one month of enrollment)
5. Current supplementation with FS or soy derivatives or allergies to them
6. Active or prior ingestion of Vitamin E exceeding 30 IU within 21 days
7. Significant liver disease (cirrhosis)
8. Significant renal dysfunction (GFR below 50 ml/hr/m2)
9. Poorly controlled diabetes (evidenced by HgbA1c>7.5% or consistently with blood glucose >250 mg/dl)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with side effects secondary to flaxseed ingestion | one month
  10 patients with cystic fibrosis were asked to consume 40 grams daily of finely ground flaxseed powder (however they wished) for one month. To assess side effects, each patient kept a journal to ascertain what side effects (if any) were most common among consumers of this dose of flaxseed. Side effects could include, but were not limited to, nausea, bloating, diarrhea or constipation. Other even rarer side effects could be bleeding, flushing, or anaphylaxis.

SECONDARY OUTCOMES:
Measure levels of flaxseed metabolism in the blood of patients with cystic fibrosis | one month
  10 patients with cystic fibrosis consumed 40 grams of flaxseed daily. One time per week (four times total), blood was drawn to assess systemic levels of flaxseed metabolites.
Measure biomarkers of systemic oxidative stress | one month
  10 patients with CF who had consumed 40 grams daily of flaxseed had urine and blood collected once weekly to ascertain potential effects of flaxseed consumption on systemic biomarkers of oxidative stress, including F2-isoprostanes, 8-oxo-dGuo, TNFa, IL-6, IFNg.

CONTACTS AND LOCATIONS:
Overall Officials: Jason B Turowski, MD, Principal Investigator — University of Pennsylvania; Denis Hadjiliadis, MD, Principal Investigator — University of Pennsylvania; Melpo Christofidou-Solomidou, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] J. B. Turowski, M. Christofidou-Solomidou, J. A. Lawson, D. Hadjiliadis, Am J Respir Crit Care Med 187;2013:A2069 Modulation Of Inflammatory And Oxidative Stress Biomarkers In Cystic Fibrosis Patients By A Dietary Botanical A94 THERAPEUTIC AND DIAGNOSTIC ADVANCES IN CYSTIC FIBROSIS / Mini Symposium / Sunday, May 19/2:00 PM-4:30 PM / Room 204 A-B (200 Level) Pennsylvania Convention Center
- [Derived] Turowski JB, Pietrofesa RA, Lawson JA, Christofidou-Solomidou M, Hadjiliadis D. Flaxseed modulates inflammatory and oxidative stress biomarkers in cystic fibrosis: a pilot study. BMC Complement Altern Med. 2015 May 13;15:148. doi: 10.1186/s12906-015-0651-2. PMID 25963404